CLINICAL TRIAL: NCT04028570
Title: A Feasibility Study Evaluating Surgery for Mesothelioma After Radiation Therapy Using Extensive Pleural Resection
Acronym: SMARTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-5987
Record Dates: First submitted 2019-04-03; First posted 2019-07-22 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Mesothelioma; Lung
Keywords: Radiation; Boost Radiation Therapy; Background Radiation Therapy; Surgery; Extensive Pleural Resection
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Intervention Model Description: 3+3 radiation dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation (Experimental): This study involves a 3+3 design. The starting cohort (n=3) will receive a neoadjuvant Background dose to the affected hemithorax (starting at 0 cGy) as well as concomitant Boost dose (of at least 2100 cGy) to a part of the gross tumour volume (GTV). The radiation will be delivered over 3 alternate days over 5-7 calendar days followed by macroscopically complete extensive pleural resection (either extra-pleural pneumonectomy or extended pleurectomy decortication, at the surgeon's discretion) after 7 to 14 days. If no dose limiting toxicities (DLTs) seen, then the Background RT dose will be increased by 600 cGy (up to 1800 cGy) and the cohort (n=3) for the next dose level will be accrued. If only 1 DLT seen, then an additional 3 patients will be treated on this dose level. If 2 or more DLTs seen at any given dose level, then the previous dose level will be defined as the maximum tolerated dose (MTD). Patients will be stratified by type of resection.
  Interventions: Radiation: Varying Doses of Background and Boost RT

INTERVENTIONS:
Radiation: Varying Doses of Background and Boost RT — 3+3 radiation dose escalation model to see the maximum tolerated dose for background and boost radiation therapy.

SUMMARY:
This study aims to find the maximum tolerated dose level for malignant pleural mesothelioma patients receiving background radiation + boost radiation, and surgery. Boost radiation is an experimental form of radiation that involves targeting non-uniform high doses of radiation to bulky pleural masses. We hypothesize the immunologic abscopal effect is an important component in controlling disease, and may be stimulated with highly hypofractionated doses. Doses will increase with every three patients who will be enrolled in the study until the background radiation reaches 1800 cGy or the maximum tolerated dose, whichever is lower.

DETAILED DESCRIPTION:
This study aims to find the maximum tolerated dose level for mesothelioma patients receiving background radiation + boost radiation, and surgery. 3 patients will start with a background radiation therapy (RT) dose of 0 cGy, and boost RT of at least 2100 cGy. If the radiation is manageable (radiation related AEs grade < 4), the next set of 3 patients will be enrolled, and the background radiation dose will be increased by 600 cGy. This will continue until the background radiation dose reaches 1800 cGy. If 1 patient exhibits dose limiting toxicities (AEs grade 4 & 5), the dose level will repeat with the next 3 patients. If 2 or more patients exhibit DLTs, the previous dose level will be determined as the maximum tolerated dose level. Surgery will be scheduled to occur approximately 1-2 weeks after completing radiation therapy, and will subsequently be followed up as per study schedule.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Good pulmonary function precluding radiation therapy (FEV1>1 L or >40% predicted or DLCO >45% predicted)
* Any patient with a new histological diagnosis of malignant pleural mesothelioma (MPM). Sarcomatoid or biphasic histologies can be included but will be analyzed separately due to their poor prognosis.
* Stage T1-3 N0-1 M0 according to the 8th edition of the tumor, node, and metastases (TNM) staging system based on conventional investigations and tests (Appendix 1). Note that the updated TNM staging system now categorizes ipsilateral mediastinal nodes as N1 disease.
* Suitable for combined modality therapy
* Informed consent.

Exclusion Criteria:

* Age < 18 years.
* Contralateral mediastinal nodal disease (N2)
* Distant metastatic disease (M1).
* Poor performance status ECOG 3-4.
* Poor pulmonary function precluding radiation therapy (FEV1<1 L or <40% predicted or diffusion lung capacity for carbon monoxide (DLCO) <45% predicted)
* Failure to provide informed consent.
* Previous thoracic irradiation.
* Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment.
* Previous chemotherapy for this or concurrent malignancy.
* Previous or concomitant malignancies except for patients with non-melanoma skin cancer, contralateral non-invasive breast cancer, prostate cancer treated with curative intent or carcinoma in situ of any other site. In addition, patients with invasive cancers treated more than 3 years previously and without evidence of recurrence will be eligible.
* Women who are currently pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose for Background Radiation | Up to five years
  AEs will be graded by CTCAE. Maximum tolerated dose is the dose level that do not result in fatal lung injury (grade 5 lung toxicity) or life-threatening or fatal treatment related toxicity (grade 4+).

SECONDARY OUTCOMES:
Patient Morbidity | Up to five years
  NCI common toxicity scale
Local recurrence | Up to five years
  Documented radiographically
Patients' quality of life | Up to five years
  Short Form Health Survey-36 (SF-36) Form
Evaluating patients' pain | Up to five years
  Assess by using the Short Form (BPI-SF)
Evaluating patients' pain | Up to five years
  Assess by using The Hospital Anxiety and Depression Scale (HADS)
Evaluating patients' pain | Up to five years
  Assess by using the EuroQol EQ-5D-5L Questionnaire
Evaluating patients' pain | Up to five years
  Assess by using the Sensitivity to Pain Traumatization Scale (SPTS)
Evaluating patients' pain | Up to five years
  Assess by using the ID Pain form
Evaluating patients' pain | Up to five years
  Assess by using the Pain Catastrophizing Scale (PCS)
Evaluating patients' pain | Up to five years
  Assess by using the Post-traumatic Stress Disorder Checklist-Civilian version (PCL-C)
Evaluating patients' pain | Up to five years
  Assess by using a variety of standard instruments including the Injustice Experience Questionnaire (IEQ).

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, PhD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No